CLINICAL TRIAL: NCT02293291
Title: Thermal Clinic Treatment in Gulf War Illness
Acronym: TCTGWI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: American Society Of Thermalism And Climatology Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GWI-2014
Record Dates: First submitted 2014-11-07; First posted 2014-11-18 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Gulf war illness
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium Water (Active Comparator): To empirically test the effects of Lithium water in violence prevention program on rates of violent attitudes and behavioral inclinations in populations whose drinking water supplies contain little or no lithium.
  To utilize an experimental design to establish statistical support for the impact of community habits related variables (protective factors) on violent attitudes and behavioral inclinations among at-risk communities To demonstrate the effect of drinking water variables (protective factors) to existing evidence-based factors (risk factors) that have proven effective in reducing violence based on previous research.
  Interventions: Dietary Supplement: Lithium Water
- MIneral water (Placebo Comparator): To empirically test the effects of Lithium water in violence prevention program on rates of violent attitudes and behavioral inclinations in populations whose drinking water supplies contain little or no lithium.
  To utilize an experimental design to establish statistical support for the impact of community habits related variables (protective factors) on violent attitudes and behavioral inclinations among at-risk communities To demonstrate the effect of drinking water variables (protective factors) to existing evidence-based factors (risk factors) that have proven effective in reducing violence based on previous research.
  Interventions: Dietary Supplement: Lithium Water

INTERVENTIONS:
Dietary Supplement: Lithium Water — To empirically test the effects of Lithium water in violence prevention program on rates of violent attitudes and behavioral inclinations in populations whose drinking water supplies contain little or no lithium.
  To utilize an experimental design to establish statistical support for the impact of community habits related variables (protective factors) on violent attitudes and behavioral inclinations among at-risk communities To demonstrate the effect of drinking water variables (protective factors) to existing evidence-based factors (risk factors) that have proven effective in GWI
  Other Names: LIWA

SUMMARY:
Although thermal therapy has been utilized in the rehabilitation of war veterans since the Roman Empire, no investigations actually exist about the use of thermal therapy in GWI, This due to the fact that nobody knows that the cure for the syndrome in GWI veterans may exist in thermal therapy which is the primary objective of this investigation.

DETAILED DESCRIPTION:
Gulf War illness (GWI) refers to the complex of symptoms that affects veterans of the 1990-1991 Gulf War at significantly excess rates. It is characterized by multiple diverse symptoms not explained by established medical diagnoses or standard laboratory tests, symptoms that typically include a combination of memory and concentration problems, persistent headache, unexplained fatigue, and widespread pain, and can also include chronic digestive difficulties, respiratory symptoms, and skin rashes. A similar profile of excess symptoms has been described in every study of U.S. Gulf War veterans from different regions and units, and in Gulf War veterans from the United Kingdom and other allied countries.

Gulf War illness is not the only health condition related to Gulf War service, but it is by far the most common. Gulf War illness prevalence estimates vary with the specific case definition used. Studies consistently indicate, however, that an excess of 25 to 32 percent of veterans who served in the 1990-1991 Gulf War are affected by a complex of multiple symptoms, variously defined, over and above rates in contemporary military personnel who did not deploy to the Gulf War. That means that between 175,000 and 210,000 of the nearly 700,000 U.S. veterans who served in the 1990-1991 Gulf War suffer from this persistent pattern of symptoms as a result of their wartime service.

Research has not supported early speculation that Gulf War illness is a stress-related condition. Large population-based studies of Gulf War veterans consistently indicate that Gulf War illness is not the result of combat or other deployment stressors, and that rates of posttraumatic stress disorder (PTSD) and other psychiatric conditions are relatively low in Gulf War veterans. Gulf War illness differs fundamentally from trauma and stress-related syndromes that have been described after other wars. No Gulf War illness-type problem, that is, no widespread symptomatic illness not explained by medical or psychiatric diagnoses, has been reported in veterans who served in Bosnia in the 1990s or in current conflicts in Iraq and Afghanistan.

Epidemiologic studies indicate that rates of Gulf War illness vary in different subgroups of Gulf War veterans. Gulf War illness affects veterans who served in the Army and Marines at higher rates than those in the Navy and Air Force, and enlisted personnel more than officers. Studies also indicate that Gulf War illness rates differ according to where veterans were located during deployment, with highest rates among troops who served in forward areas. More specifically, studies consistently show that the rate of Gulf War illness is associated with particular exposures that veterans encountered during deployment.

Identified links between veteran-reported exposures and Gulf War illness have raised a great deal of interest, but have also been the source of considerable confusion. The use of self-reported exposure information raises a number of concerns, most obviously in relation to recall bias. These concerns emphasize the importance of assessing findings across a broad spectrum of studies, rather than relying on results from individual studies, and of evaluating the impact of recall and other information bias on study results where possible.

Approximately 34-65% of Gulf War veterans (GWV) continue to suffer from chronic multi symptom illness (CMI).Novel pharmacological treatment approaches are needed to improve the health of these veterans. The current study aims to target neurological alterations that have been described in veterans of the 1991Gulf War. In particular, a low lithium has been associated with Gulf War deployment and symptoms of CMI. A correct Lithium level trough of dietary supplement and external bath have effects on multiple systems, including the immune system, autonomic nervous system, and the central nervous system, this system is a potential target of treatment in CMI To be a factor in the multifactorial development of GWI, the American Society of Thermalism and Climatology has reviewed each of the aggressive external factors that the investigators veterans have been exposed to during their deployment in the Gulf and the symptoms this exposure may cause.

After six months of study the investigators have concluded that the syndrome is a multi-systematic response to multiple factors so the treatment must be multiple therapeutic treatment. If the ones the investigators treat are man-nature unbalanced, the cure is to be found in the balance so climatological hydro therapy is the first source to achieve this balance (TA Silega theory).

Although thermal therapy has been utilized in the rehabilitation of war veterans since the Roman Empire, no investigations actually exist about the use of thermal therapy in war veterans with the knowledge that the cure for the syndrome in GWI veterans may exist in thermal therapy which is the primary objective of this investigation.

Using data for the last 3 year for New York metropolitan VA office (2011-2013), will show that' the incidence rates of GWI are significantly higher in these veterans whose plasma contain a unbalance of electrolytes in special lithium than in veterans with normal electrolytes levels ranging.

These results will suggest that lithium has moderating effects on suicidal and violent criminal behavior at levels that may be encountered in GWI. Comparisons of lithium levels in the respective veterans, with the incidences GWI from 2011-2013 also will produced statistically significant inverse associations, whereas consistent associations will observed with the reported GWI. These results will suggest that lithium at low dosage levels has a generally beneficial effect on human behavior, which may be associated with the functions of lithium as a nutritionally-essential trace element. Subject to confirmation by controlled experiments with high-risk military populations, increasing the human lithium intakes by supplementation, or the lithiation of drinking water in military bases campuses is suggested as a possible means of GWI reduction at the individual and community level.

Lithium is a trace element that appears to be essential for higher animals (1, 2). However, although the element is widely used at pharmacological dosages in the treatment of various mental disorders (3), its effects at normal nutritional levels have not yet received much attention. Dawson, Moore and McGanity (4) previously compared the lithium concentrations in the regional drinking water supplies with the incidence of admissions and readmissions for psychoses, neuroses, and personality disorders in Texas state mental hospitals and observed a statistically significant inverse relationship. The same authors subsequently showed that the homicide rates were also inversely correlated with the lithium levels in the drinking water and the urinary excretion of lithium by normal residents in their respective areas (5). The associations remained significant after consideration of possible confounding variables, such as population density, the distance to the nearest state hospitals, and rainfall. Although rainfall was positively correlated with the county rates of first mental hospital admission, as well as with homicide rates, rainfall was also found to be inversely correlated with the lithium levels in the drinking water and the urinary excretion of lithium by healthy subjects, demonstrating a dilution effect of rainfall on the water supplies. With the suicide rates, the association with water lithium levels was inverse, but did not reach statistical significance. Since incidence data for only two years, 1967-1969, were used in these studies, the investigators decided to reinvestigate the relationships between drinking water lithium with homicide and suicide rates for 10 years, using data from 1978-1987, and extend the study to other GWIs (rapes, robberies, thefts, burglaries, assault, motor vehicle theft, and the total GWI rate). As the addiction to narcotics may be regarded as a self-destructive trait, which thus could depend on the same environmental influences as suicide, comparisons were also made between the drinking water lithium levels in the respective veterans and the incidences of arrests for possession of opium, cocaine, and their derivatives (morphine, heroin, and codeine), and possession of marijuana, as well as arrests for drunk driving and using data from 2011-201 This research will suggest a beneficial effect of lithium at GWI. These could be related to the roles of lithium as an essential trace element.

Lithium as the carbonate at therapeutic dosage (300 mg/d) has previously been used to control episodic outbreaks of rage among prisoners (10, 11) and in the management of drug abusers (12). Animal experiments have demonstrated that lithium suppresses the cocaine-induced super- sensitivity, as well as the super sensitivity induced by haloperidol, the kindling phenomenon following the chronic application of pentylene-tetrazole, a central nervous system stimulant, and head-twitching in response to the administration of mescaline (13). Furthermore, lithium has been found to decrease distractibility by irrelevant stimuli and produce a dose-independent improvement of selective attention to stimuli that provide detailed information about the environment. It prevents behavioral alterations owing to social isolation, lowers aggressively owing to confinement in isolated environments, and causes a normalization of spontaneous motor activity (14). The majority of these effects may be associated with the dampening of phosphoinositide-mediated neuro- transmission, which was also suggested to explain the normalizing effects of lithium in treating both mania and depression (15).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are primarily diagnosed with PTSD (Posttraumatic Stress Disorder: 309.81) using DSM-IV-TR criteria. The CAPS-DX (Clinician-Administered PTSD Scale-DX) and M.I.N.I. (The Mini International Neuropsychiatric Interview, Japanese version 5.0.0. [2003]) will be used for diagnosis
* Patients aged 18 and <65 at the time of signing the Informed consent
* Male and female patients
* Inpatient/outpatient status: Both are permitted
* Patients who are able to give written informed consent in person (i.e., patients who are capable of giving written informed consent on their own)
* Patients whose combined score of the CAPS-SX standard B, C, and D is over 50

Exclusion Criteria:

* Patients primarily diagnosed with a DSM-IV-TR Axis I disorder other than PTSD (e.g. major depressive disorder, dysthymic disorder, specific phobia [simple phobia], obsessive-compulsive disorder, panic disorder, etc.) within 6 months of week -4 (start of baseline phase)
* Patients presenting with a current major depressive episode that preceded the diagnosis of PTSD
* Patients who are pregnant, lactating or of childbearing potential and are likely to become pregnant
* Patients receiving another investigational product within 12 weeks before Week -4 (start of baseline phase)
* Patients with a history or complication of manic psychosis
* Patients with a history or complication of convulsive disorder (epilepsy, etc.)
* Patients with a diagnosis or complication of a cognitive disorder (MMSE <=24 points)
* Patients with a history and complication of serious cerebral organic disorder. (e.g. cerebrovascular disorder, meningitis, degenerative disease and other neurological disorders and seizures; however, bleeding in the upper arachnoid membrane should not be excluded)
* Patients unable or unwilling to undergo the fMRI procedure (e.g., cerebrovascular clipping surgery, pacemaker, any internal metals with magnetism, and claustrophobia)
* Patients with glaucoma
* Patients with a known tendency for bleeding or those with predisposing conditions
* Patients with serious physical symptoms (cardiac, hepatic and renal dysfunction, or hematopoietic dysfunction, etc.). For seriousness, Grade 3 of "Criteria for seriousness of adverse reactions to drugs, etc. (Yakuan No.80)" is used as an index
* Patients with a history or complication of cancer or malignant tumour
* Patients with chronic hepatitis type B and/or C which is positive of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibody
* Others whom the investigator or sub-investigator considers ineligible for or unable to participate in the investigation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Number of veterans (GWI) with positive response to lithium water therapy | 52 weeks
  General response to Lithium water therapy in veterans from Gulf War

CONTACTS AND LOCATIONS:
Overall Officials: Garis Silega, MD, Principal Investigator — America Society of thermalism
Locations (1):
- Gaviota Clinic, Newark, New Jersey, United States